CLINICAL TRIAL: NCT04450784
Title: ObServatory Children Acute RElated Therapy Leukemia
Acronym: OSCARE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/31
Record Dates: First submitted 2020-06-09; First posted 2020-06-30 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Secondary; Acute myeloid Leukemia; Children
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Secondary Acute Myeloid Leukemias (AML) of the child
  Interventions: Other: collection of the clinical and biological characteristics of secondary AMLs in children

INTERVENTIONS:
Other: collection of the clinical and biological characteristics of secondary AMLs in children — to record scientific and medical information on cases of secondary Acute Myeloid Leukemias that have occurred in France since 2013

SUMMARY:
Acute Myeloid Leukemias (AML) of the child are a rare disease and its prognosis varies according to the subgroup. Secondary AMLs remain a subgroup of poor prognosis, whose cytogenetic and molecular characteristics and prognostic value differ in part from de novo AMLs. The purpose of this national observatory is to record scientific and medical information on cases of secondary AML that have occurred in France since 2013 in order to improve the treatment of children and adolescents with this disease in the years to come. This national observatory will contribute to better knowledge and progress in research into these diseases.

DETAILED DESCRIPTION:
Therapy-related myeloid neoplasms (t-MNs) are a group of hematologic diseases that arise after chemotherapy and/or radiation therapy for a previous cancer or rarely autoimmune diseases. t-MNs had been included in the group of AMLs and remain as a distinct category also in the recent 2016 revision of the WHO classification of myeloid neoplasm and acute leukemia. The latency between exposition to anticancer drugs and development of t-MN may vary from some months up to 10 years, even considering the age at diagnosis of the primary malignancy, the kind of cytotoxic treatment previously used, and the cumulative dose and dose intensity. The prognosis of s-AML is generally considered to be poorer than that of de novo AML. The disease tends to be refractory to chemotherapy, and patients' tolerance of treatment generally is reduced because of prior therapies. 5-year event-free survival (EFS) and overall survival (OS) rates of pediatric t-AML/t-MDS have been reported to be 14% to 30%. However, the results are conflicting and overall lacking when compared with those in adults. The purpose of this national observatory is to record scientific and medical information on cases of secondary Acute Myeloid Leukemias that have occurred in France since 2013 in order to improve the treatment of children and adolescents with this disease in the years to come. The primary objective is to evaluate the association of potential prognostic factors (including clinical-biological factors) with the overall survival of children and adolescents aged 0-18 years diagnosed with secondary AML. The secondary objectives are to test the feasibility of setting up a French national database of secondary AMLs for children and adolescents as a first step towards European implementation, to assess the association of potential prognostic factors with event free survival and the occurrence of treatment-related toxicities, to characterize the molecular abnormalities associated with secondary AMLs in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-18 years
* Patient with first cancer
* Diagnosis of secondary AML
* Patients treated in a SFCE (Société française des cancers de l'enfant) center
* For cases included in the prospective from March 2019 onwards: Consent of holders of parental authority and consent of the child of understanding age

Exclusion Criteria: None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents aged 0-18 years diagnosed with secondary AML
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
potential clinical-biological prognostic factors - patient characterics | through study completion, an average of 6 months
  patient characteristics are sex, patient's age at the start of treatment for secondary AML, date of birth, personal history of genetic predisposition (including brittle diseases - see below), family history of cancers (1st or 2nd degree)
potential clinical-biological prognostic factors - first cancer characteristics | through study completion, an average of 6 months after patient inclusion
  First cancer characteristics are age of onset, determined from the date of diagnosis, and histology, determined by anatomo-pathological diagnosis.
potential clinical-biological prognostic factors :first cancer treatment : types of treatments received | through study completion, an average of 6 months after patient inclusion
  type of treatment: chemotherapy (Anthracyclines, Alkylating agents) and / or radiotherapy and/or Marrow autograft or allograft
potential clinical-biological prognostic factors - first cancer treatments: response to treatment | through study completion, an average of 6 months after patient inclusion
  response measured by bone marrow assessment using morphology and minimal residual disease (MRD) assessment : no response, partial response, complete remission
potential clinical-biological prognostic factors - first cancer treatments: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 6 months after patient inclusion
  nature, incidence and severity of adverse events (AEs)
potential clinical-biological prognostic factors - first cancer treatments: duration of treatment | through study completion, an average of 6 months after patient inclusion
  duration of treatment determined from the start and end dates
potential clinical-biological prognostic factors - first cancer treatments: cumulative dose received | through study completion, an average of 6 months after patient inclusion
  cumulative dose of each type of treatment received ( chemotherapy (Anthracyclines, Alkylating agents) and / or radiotherapy and/or Marrow autograft or allograft)
potential clinical-biological prognostic factors - secondary AML characteristics: date of diagnosis | through study completion, an average of 6 months after patient inclusion
  date of diagnosis
potential clinical-biological prognostic factors - secondary AML characteristics: median time of onset compared to the date of end of treatment for the 1st cancer | through study completion, an average of 6 months after patient inclusion
  median time of onset compared to the date of end of treatment for the 1st cancer
potential clinical-biological prognostic factors - secondary AML characteristics : hematological data assessed by morphology | through study completion, an average of 6 months after patient inclusion
  Leukocytes at diagnosis of secondary AML (G/L)
potential clinical-biological prognostic factors - secondary AML characteristics: cytogenetic data | through study completion, an average of 6 months after patient inclusion
  karyotype, exclusive and cumulative anomalies
potential clinical-biological prognostic factors - secondary AML characteristics: molecular data | through study completion, an average of 6 months after patient inclusion
  molecular data assessed by Next-Generation Sequencing panel
potential clinical-biological prognostic factors - secondary AML treatment: duration of treatment | through study completion, an average of 6 months after patient inclusion
  duration of treatment determined from the start and end dates
potential clinical-biological prognostic factors - secondary AML treatment: type of treatment | through study completion, an average of 6 months after patient inclusion
  chemotherapy received and bone marrow transplantation
potential clinical-biological prognostic factors - secondary AML treatment : response to treatment | through study completion, an average of 6 months after patient inclusion
  response measured by bone marrow assessment using morphology and minimal residual disease (MRD) assessment : no response, partial response, complete remission
potential clinical-biological prognostic factors - secondary AML treatment: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 6 months after patient inclusion
  nature, incidence and severity of adverse events (AEs)
potential clinical-biological prognostic factors - Overall Survival (OS) | at the end of the 2 years of the inclusion period
  Evaluated as time from diagnostic of the second AML to death from any cause or date last seen for patients who are alive at the end of the trial

SECONDARY OUTCOMES:
feasibility of setting up a French national database of secondary AMLs for children and adolescents - Number of cases included over the period | at the end of the 2 years of the inclusion period
  Number of cases included over the period
feasibility of setting up a French national database of secondary AMLs for children and adolescents - Missing Data | at the end of the 2 years of the inclusion period
  Proportion and type of missing data in the database after the base freeze
feasibility of setting up a French national database of secondary AMLs for children and adolescents - Centre participation rates | at the end of the 2 years of the inclusion period
  Centre participation rates
association of potential prognostic factors with event free survival and the occurrence of treatment-related toxicities- Recurrence of the disease | at the end of the 2 years of the inclusion period
  Recurrence of the disease : Relapse criteria (in a patient who has had complete remission):
  ≥ 5% blasts in the bone marrow (not attributable to post chemotherapy regeneration)
association of potential prognostic factors with event free survival and the occurrence of treatment-related toxicities- Treatment-related toxicities | at the end of the 2 years of the inclusion period
  Treatment-related toxicities : Metabolic / endocrine complications in particular: growth retardation, hypothyroidism, gonadal insufficiency; Organic complications, in particular: renal failure, heart failure, respiratory failure ; Graft versus host reaction (GvH)

IPD SHARING:
Plan to Share IPD: No